CLINICAL TRIAL: NCT04145960
Title: Evaluation of Prognostic Monitoring for Women Who Have Completed Standard Treatment for Breast Cancer Via Analysis of Immunoinflammation-related Protein Complexes in Blood
Brief Title: Evaluation of Prognostic Monitoring for Women Who Have Completed Standard Treatment for Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yali XU, Principal Investigator, Peking Union Medical College Hospital
Other Study IDs: PUMCH-BC500
Record Dates: First submitted 2019-08-12; First posted 2019-10-31 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — 1 mL of blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymph node metastasis: Axillary lymph node metastasis ≥ 4 Lymph nodes

SUMMARY:
The relationship between immune inflammation-related protein complexes in blood and recurrence or metastasis of breast cancer will be studied.

DETAILED DESCRIPTION:
200 patients with breast cancer will be followed up. Peripheral venous blood was collected every 3 to 6 months. Change regularity of breast cancer-specific immune inflammation-related protein complexes in blood at different follow-up time points will be studied. The relationship between disease-specific protein complexes and pathological state of patients will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Postoperative pathology confirmed invasive breast cancer after surgery for breast tumors
* Breast cancer-related chemotherapy and radiotherapy completed
* axillary lymph node metastasis ≥ 4
* age ≤ 60 years old

Exclusion Criteria:

* Male
* Aged above 60
* Breast Carcinoma in situ
* Women in pregnancy or breastfeeding
* Suffering from other malignant tumors
* Non-compliant patient

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The participant eligibility is based on the physiological sex.
Study Population: Patients with high risk of recurrence and metastasis of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
immune inflammation-related protein complexes | 2 years
  The change of immune inflammation-related protein complexes which is measured by gel permeation chromatography.
blood markers | 2 years
  The expression of CA153, CEA, CA125 in the blood of the patients, which are measured by electro-chemiluminescence immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Yali Xu, Principal Investigator
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No